CLINICAL TRIAL: NCT04249362
Title: A Phase II, Open-label, Multicenter, International Study of Durvalumab Following Radiation Therapy in Patients With Stage III, Unresectable Non-Small Cell Lung Cancer Who Are Ineligible for Chemotherapy
Brief Title: Study of Durvalumab Following Radiation Therapy in Patients With Stage 3 Unresectable NSCLC Ineligible for Chemotherapy
Acronym: DUART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4194C00009; 2019-004336-31 (EudraCT Number)
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Radiation therapy; Phase II; Palliative Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Experimental): Patients received standard radiotherapy [60 gray (Gy) ± 10% or hypofractionated BED] prior to study entry.
  Interventions: Drug: Durvalumab
- Cohort B (Experimental): Patients received palliative radiotherapy [40 to < 54 Gy or hypofractionated BED] prior to study entry.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — All patients will receive 1500 mg durvalumab via IV infusion q4w for up to a maximum of 12 months.
  Other Names: MEDI4736

SUMMARY:
This is a Phase II open-label, single-arm, multicenter, international study to evaluate the clinical activity of durvalumab in patients with Stage III unresectable NSCLC who are deemed to be ineligible for chemotherapy per Investigator assessment. Patients will be enrolled into 2 cohorts according to radiotherapy pretreatment dose (Cohort A: standard radiation therapy [60 gray (Gy) ± 10% or hypofractionated bioequivalent dose (BED)]; Cohort B: palliative radiation therapy [40 to < 54 Gy or hypofractionated BED])

DETAILED DESCRIPTION:
This is a Phase II open-label, single-arm, multicenter, international study to evaluate the clinical activity of durvalumab in patients with Stage III unresectable NSCLC who have an Eastern Cooperative Oncology Group (ECOG) PS of 0 to 2 and who were treated with radiotherapy but are ineligible for chemotherapy. Patients will be enrolled into 2 cohorts according to the dose of radiotherapy received prior to study entry (Cohort A: Standard Radiotherapy [60 Gy ± 10% or hypofractionated BED]; Cohort B: Palliative Radiotherapy [40 to < 54 Gy or hypofractionated BED]). Patients must not have progressed following radiation therapy, and radiation therapy must be completed within 6 weeks (42 days) prior to first study drug administration. The last dose of radiation therapy is defined as the day of the last radiation treatment session. All patients will receive 1500 mg durvalumab via IV infusion every 4 weeks (q4w) for up to a maximum of 12 months (up to 13 doses/cycles)

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Age ≥ 18 years at study entry.
3. Histologically or cytologically documented NSCLC with locally-advanced, unresectable Stage III disease.
4. Deemed ineligible for chemotherapy per Investigator assessment.
5. Receipt of radiation therapy that was completed within 42 days prior to first study drug administration.
6. Must have received a total dose of radiation of 40 to 66 Gy (standard or hypofractionated BED).
7. Must not have progressed following radiation therapy, as per Investigator assessed RECIST 1.1 criteria: a) Patients with measurable disease and/or nonmeasurable and/or no evidence of disease assessed at baseline by computed tomography /magnetic resonance imaging will be eligible for this study. b) Prior irradiated lesions may be considered measurable and selected as target lesions (TLs) providing they fulfill the other criteria for measurability.
8. World Health Organization/ECOG performance status of ≤2.
9. No prior exposure to immune-mediated therapy including, but not limited to, anti-CTLA-4, anti-PD-1, anti-PD-L1, and antiprogrammed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
10. Patients must have adequate organ and marrow function as defined below:

    * Hemoglobin ≥ 9.0 g/dL
    * Absolute neutrophil count ≥ 1.0 × 109 /L
    * Platelet count ≥ 75 × 109/L
    * Serum bilirubin ≤ 1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome.
    * Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × ULN
    * Measured creatinine clearance > 30 mL/min or calculated CL > 30 mL/min as determined by Cockcroft-Gault
11. Life expectancy of greater than 12 weeks.
12. Body weight greater than 30 kg at study entry and at first study drug administration

Exclusion Criteria:

1. Patients with locally-advanced NSCLC whose disease has progressed following radiation therapy.
2. Mixed small cell lung cancer and NSCLC histology.
3. History of allogeneic organ transplantation.
4. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome).
5. Uncontrolled intercurrent illness (e.g., ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris)
6. History of another primary malignancy except for (a) malignancy treated with curative intent and with no known active disease ≥ 5 years before the first study drug administration, (b) adequately treated nonmelanoma skin cancer or lentigo maligna without evidence of disease, and c) treated carcinoma in situ without evidence of disease.
7. History of leptomeningeal carcinomatosis
8. History of active primary immunodeficiency
9. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus
10. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, lymphopenia, and the laboratory values defined in the inclusion criteria
11. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
12. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab
13. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of durvalumab.
14. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
15. Participation in another clinical study with an IP administered in the last 4 weeks.
16. Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
17. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment
18. Patients who refuse chemotherapy by their own decision.
19. Involvement in the planning and/or conduct of the study
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control.
21. Judgment by the Investigator that the patient should not participate in the study
22. Genetics research study (optional):

Exclusion criteria for participation in the optional genetics research component of the study include: a) Previous allogeneic bone marrow transplant b)Nonleukocyte-depleted whole blood transfusion within 120 days of genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Andrea Riccardo Filippi, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (34):
- United States (3):
  - Research Site, Tucson, Arizona
  - Research Site, Tampa, Florida
  - Research Site, Royal Oak, Michigan
- France (5):
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Rouen
- Italy (12):
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Modena
  - Research Site, Monza
  - Research Site, Negrar
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Roma
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Olsztyn
  - Research Site, Szczecin
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Sabadell(Barcelona)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Filippi AR, Dziadziuszko R, Garcia Campelo MR, Paoli JB, Sawyer W, Diaz Perez IE. DUART: durvalumab after radiotherapy in patients with unresectable, stage III NSCLC who are ineligible for chemotherapy. Future Oncol. 2021 Dec;17(34):4657-4663. doi: 10.2217/fon-2021-0952. Epub 2021 Nov 15. PMID 34775804
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00009&attachmentIdentifier=dc99eaef-457a-4ade-b223-4e5ae1f63416&fileName=246839_CSP_Final_Draft__PDFA_Redacted.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00009&attachmentIdentifier=5ed542aa-f1fc-42ab-b28e-5b4e5e0eb29e&fileName=246839_SAP_Final_Draft__PDFA_Redacted.pdf&versionIdentifier=
- See also: CSR synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00009&attachmentIdentifier=589ee75a-0203-44f6-9623-a75377cf7c8c&fileName=246839_PA_CSR_synopsis_Final_Draft__PDFA_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled and received study treatment at 29 sites in 5 countries (France, Italy, Poland, Russian Federation, and Spain). The data in this report are based on study start date (first patient enrolled: 26 November 2020 till final analyses data cut-off date of 06 December 2023.
Pre-assignment Details: Eligible patients who met all inclusion criteria were enrolled in the study. However, one patient was later found to have an important protocol deviation, and many other patients had protocol deviations. Study assessments followed scheduled timeline. Enrolled patients had Stage III unresectable Non-Small Cell Lung Cancer (NSCLC), an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2, had been treated with radiotherapy, and were ineligible for chemotherapy.
Groups:
- Durvalumab Cohort A: Standard Radiotherapy (RT): Patients who received standard RT [60 gray (GY) ± 10% or hypofractionated bioequivalent dose (BED)] before study entry were administered a fixed dose of 1500 mg of durvalumab via intravenous (IV) infusion every 4 weeks (q4w) for a duration of 12 months (up to 13 doses/cycles), or until clinical progression or radiological progression defined by the response evaluation criteria in solid tumors version (RECIST 1.1), unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Durvaumab Cohort B: Palliative Radiotherapy (RT): Patients who received palliative RT [40 to < 54 Gy or hypofractionated BED] before study entry were administered a fixed dose of 1500 mg of durvalumab via IV infusion q4w for a duration of 12 months (up to 13 doses/cycles), or until clinical progression or radiological progression defined by the RECIST 1.1, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT)
Started | 53 | 49
Completed | 53 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.7 (9.18) | 78.8 (6.71) | 76.7 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 38 | 35 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 45 | 91
  Other | 1 | 0 | 1
  Unknown | 3 | 1 | 4
  Missing | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 45 | 43 | 88
  Missing | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3 and Grade 4 Possibly-related Adverse Events (PRAEs)
Description: The safety and tolerability profile of durvalumab as defined by Grade 3 and Grade 4 PRAEs within 6 months from the initiation of durvalumab treatment. A PRAE was any TEAE with a possible relatedness to durvalumab, or where the relatedness was missing. If relatedness of a TEAE was missing at the primary DCO (30 March 2023) the TEAE was considered a PRAE.
Time Frame: From first dose of durvalumab treatment until 6 months after initiation of durvalumab treatment
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab Total: Patients who received standard RT [60 gray (GY) ± 10% or hypofractionated BED)] or palliative RT [40 to < 54 Gy or hypofractionated BED] before study entry were administered a fixed dose of 1500 mg of durvalumab via IV infusion q4w for a duration of 12 months (up to 13 doses/cycles), or until clinical progression or radiological progression defined by the RECIST 1.1, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Participants | 5 | 5 | 10

2. Secondary Outcome: Median Progression-free Survival (mPFS)
Description: Progression-free survival is defined as the time from the date of first dose of durvalumab until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient discontinues durvalumab or receives another anticancer therapy prior to progression according to RECIST 1.1 as assessed by the Investigator. Patients who had not progressed or died at the time of analysis were censored at the date of their last evaluable tumor assessment. If a patient progressed or died after two or more missed visits, they were censored at the date of the latest evaluable assessment prior to the missed visits.
Time Frame: From the first date of treatment until the date of objective disease progression or death or data cut-off date (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Months | 10.3 [7.49 to 16.56] | 7.6 [5.55 to 11.04] | 9.2 [7.39 to 11.93]

3. Secondary Outcome: Progression-free Survival at 6 Months (PFS6)
Description: as for outcome 2
Time Frame: From the first date of treatment until the date of objective disease progression or death (6 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Percentage of patients | 67.1 [51.96 to 78.43] | 59.3 [43.38 to 72.07] | 63.3 [52.62 to 72.25]

4. Secondary Outcome: Progression-free Survival at 12 Months (PFS12)
Description: as for outcome 2
Time Frame: From the first date of treatment until the date of objective disease progression or death (12 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Percentage of patients | 46.8 [31.88 to 60.36] | 31.8 [18.13 to 46.32] | 39.6 [29.28 to 49.76]

5. Secondary Outcome: Median Overall Survival (mOS)
Description: The OS is defined as the time from the date of first dose of durvalumab until death due to any cause. Patients who were not known to have died at the time of analysis were censored at the last recorded date when they were known to have been alive.
Time Frame: From the first date of treatment until death or data cut-off due to any cause (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Months | 21.1 [11.60 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events. | 16.8 [10.64 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events. | 21.1 [14.75 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events.

6. Secondary Outcome: Overall Survival at 12 Months (OS12)
Description: as for outcome 5
Time Frame: From the first date of treatment until death due to any cause (12 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Percentage of patients | 64.0 [49.01 to 75.58] | 65.5 [49.87 to 77.26] | 64.7 [54.21 to 73.34]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the proportion (%) of patients with an overall response of complete response (CR) or partial response (PR) (confirmed by a follow-up scan at least 4 weeks after showing CR or PR) per RECIST 1.1 criteria. CR is disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to < 10 mm. PR is at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: From 8 weeks ±1 week after durvalumab treatment initiation and continue every 8 weeks (q8w) ±1 week through 48 weeks and every 12 weeks (q12w) ±1 week until disease progression or data cut-off (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Percentage of patients | 34.0 [21.5 to 48.3] | 24.5 [13.3 to 38.9] | 29.4 [20.8 to 39.3]

8. Secondary Outcome: Duration of Response (DoR)
Description: The DoR is defined as the time from the date of first documented response (which is subsequently confirmed) until the first date of documented progression per RECIST1.1 or death in the absence of disease progression.
Time Frame: as for outcome 7
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment. Number of participants analyzed and number analyzed here represents number of patients with objective response.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 18 | 12 | 30
Weeks | 56.9 [31.00 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events. | 34.1 [24.29 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events. | 56.9 [31.14 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events.

9. Secondary Outcome: Lung Cancer Mortality
Description: The lung cancer mortality (NSCLC-related death) is assessed using the deaths which are reported as 'NSCLC-related' and is defined as the time (days) from the date of first dose of durvalumab until date of death due to lung cancer.
Time Frame: From date of treatment start until death due to lung cancer (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Months | 30.9 [16.92 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events. | NA [14.75 to NA] — Median and upper limit of CI is not calculable due to insufficient number of patients with events. | 30.9 [16.82 to NA] — Upper limit of CI is not calculable due to insufficient number of patients with events.

10. Secondary Outcome: Number of Patients With Events (AEs)
Description: The safety and tolerability profile of durvalumab treatment, including all adverse events (AEs) was assessed.
Time Frame: From screening (Day -28) till data cut-off (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Participants
  Any AE | 50 | 49 | 99
  Any PRAE (Investigator-assessed [IA]) | 31 | 31 | 62
  Any AE of CTCAE Grade 3 or Grade 4 | 20 | 21 | 41
  Any AE of CTCAE Grade 3 or Grade 4, possibly related to durvalumab treatment (IA) | 6 | 5 | 11
  Any AE with outcome of death | 5 | 2 | 7
  Any AE with outcome of death, possibly related to treatment (IA) | 1 | 0 | 1
  Any SAE (including events with outcome of death) | 23 | 18 | 41
  Any SAE (including events with outcome of death), possibly related to treatment (IA) | 5 | 3 | 8
  Any AE leading to discontinuation of treatment | 13 | 9 | 22
  Any AE leading to discontinuation of treatment, possibly related to treatment (IA) | 7 | 5 | 12
  Any AE leading to treatment interruption | 25 | 23 | 48
  Any AE leading to treatment interruption, possibly related to treatment | 6 | 7 | 13
  Any AESI (including events with outcome of death) (IA) | 25 | 21 | 46
  Any AESI (including events with outcome of death), possibly related to treatment (IA) | 19 | 14 | 33
  Any Adverse event of potential interest (AEPI) (including events with outcome of death) (IA) | 21 | 22 | 43
  Any AEPI (including events with outcome of death), possibly related to treatment (IA) | 14 | 15 | 29
  Any imAE (IA) | 27 | 24 | 51
  Any imAE, possibly related to treatment (IA) | 26 | 24 | 50

11. Secondary Outcome: Number of Patients With Adverse Events of Special Interests (AESIs)
Description: The safety and tolerability profile of durvalumab treatment, including all adverse events (AEs) was assessed. An AESI is an AE of scientific and medical interest specific to the understanding of durvalumab. AESIs for durvalumab include, but are not limited to, events with a potential inflammatory or immune-mediated mechanism and which may require more frequent monitoring and/or interventions such as steroids, immunosuppressants and/or hormone replacement therapy. Here, number of patients experienced AESIs are presented. Serious adverse event of special interests (SAESIs).
Time Frame: From screening (Day -28) till data cut-off (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Participants
  Any AESIs | 25 | 21 | 46
  Any AESIs of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 | 4 | 1 | 5
  Any SAESIs [including events with outcome = death]) | 4 | 1 | 5
  Any AESIs with outcome = death | 1 | 0 | 1
  Any AESIs, causally related to treatment | 19 | 14 | 33
  Any AESIs of CTCAE Grade 3 or 4, causally related to treatment | 4 | 1 | 5
  Any SAESIs, causally related to treatment | 4 | 1 | 5
  Any AESIs with outcome = death, causally related to treatment | 1 | 0 | 1
  AESIs: Received systemic corticosteroids | 5 | 8 | 13
  AESIs: Received high dose steroids | 4 | 6 | 10
  AESIs: Received endocrine therapy | 6 | 5 | 11
  AESIs: Received other immunosuppressants | 0 | 0 | 0
  Any AESIs leading to discontinuation of durvalumab treatment | 4 | 3 | 7
  AESIs: Event outcome resolved | 13 | 12 | 25
  AESIs: Event outcome not resolved | 11 | 9 | 20

12. Secondary Outcome: Number of Patients With Immune-mediated Adverse Events (imAEs)
Description: The safety and tolerability profile of durvalumab treatment, including all adverse events (AEs) was assessed. An imAE is defined as an AESI that is associated with drug exposure and is consistent with an immune-mediated mechanism of action and where there is no clear alternate etiology. Here, number of patients experienced imAEs are presented. Immune-mediated serious adverse events (imSAEs)
Time Frame: From screening (Day -28) till data cut-off (36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of durvalumab treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
Number analyzed (Participants) | 53 | 49 | 102
Participants
  Any imAEs | 11 | 15 | 26
  Any imAEs of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4 | 2 | 3 | 5
  Any imSAEs [including events with outcome = death]) | 3 | 2 | 5
  Any imAEs with outcome = death | 1 | 0 | 1
  Any imAEs, causally related to treatment | 10 | 12 | 22
  Any imAEs of CTCAE Grade 3 or 4, causally related to treatment | 2 | 3 | 5
  Any imSAEs, causally related to treatment | 3 | 2 | 5
  Any imAEs with outcome = death, causally related to treatment | 1 | 0 | 1
  imAEs: Received systemic corticosteroids | 7 | 13 | 20
  imAEs: Received high dose steroids | 5 | 7 | 12
  imAEs: Received endocrine therapy | 6 | 5 | 11
  imAEs: Received other immunosuppressants | 0 | 0 | 0
  Any imAEs leading to discontinuation of durvalumab treatment | 3 | 4 | 7
  imAEs: Event outcome resolved | 5 | 8 | 13
  imAEs: Event outcome not resolved | 5 | 7 | 12

ADVERSE EVENTS:
Time Frame: From screening (Day -28) till data cut-off (36 months)
Arm/Group | Durvalumab Cohort A: Standard Radiotherapy (RT) | Durvaumab Cohort B: Palliative Radiotherapy (RT) | Durvalumab Total
All-Cause Mortality (participants affected / at risk) | 23/53 | 23/49 | 46/102
Serious Adverse Events (participants affected / at risk) | 23/53 | 18/49 | 41/102
Other Adverse Events (participants affected / at risk) | 47/53 | 45/49 | 92/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Cohort A: Standard Radiotherapy (RT) (N=53) | Durvaumab Cohort B: Palliative Radiotherapy (RT) (N=49) | Durvalumab Total (N=102)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4) | 5 (5)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 1 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Cohort A: Standard Radiotherapy (RT) (N=53) | Durvaumab Cohort B: Palliative Radiotherapy (RT) (N=49) | Durvalumab Total (N=102)
COVID-19 (Infections and infestations) | 6 (6) | 3 (3) | 9 (9)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 3 (4) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 6 (8) | 19 (22)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 2 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 5 (5) | 11 (11)
Hypothyroidism (Endocrine disorders) | 9 (9) | 6 (8) | 15 (17)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 6 (7) | 14 (15)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 6 (9)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Periorbital oedema (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 5 (5) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 12 (13) | 21 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8) | 19 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 7 (7)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 10 (12) | 13 (15)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 7 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (9) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 6 (6) | 14 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6) | 10 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 13 (14) | 8 (9) | 21 (23)
Fatigue (General disorders) | 1 (1) | 10 (10) | 11 (11)
Oedema peripheral (General disorders) | 3 (3) | 5 (5) | 8 (8)
Pyrexia (General disorders) | 8 (9) | 8 (9) | 16 (18)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (3) | 7 (7)
Amylase increased (Investigations) | 3 (3) | 2 (4) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 2 (3) | 5 (6)
Blood creatinine increased (Investigations) | 2 (2) | 4 (6) | 6 (8)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1) | 4 (4)
Blood thyroid stimulating hormone decreased (Investigations) | 2 (3) | 0 (0) | 2 (3)
Blood urea increased (Investigations) | 3 (5) | 1 (1) | 4 (6)
Blood uric acid increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
C-reactive protein increased (Investigations) | 4 (4) | 1 (1) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 2 (2) | 5 (5)
Lipase increased (Investigations) | 1 (2) | 2 (2) | 3 (4)
Neutrophil count increased (Investigations) | 4 (6) | 0 (0) | 4 (6)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT04249362/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT04249362/SAP_003.pdf